CLINICAL TRIAL: NCT03417609
Title: Interest of a Tongue Strength Measurement in the Screening for Sarcopenia in Hospitalized Elderly Patients
Status: Completed | Type: Observational
Sponsor: Murielle Surquin (Other)
Responsible Party: Sponsor-Investigator, Murielle Surquin, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-sarcopenia-tongue
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Tongue strength
MeSH Terms: conditions — Sarcopenia | interventions — Blood Specimen Collection; Absorptiometry, Photon; Walking Speed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenia: Elderly patients with sarcopenia
  Interventions: Device: Tongue strength measurement; Procedure: Blood sampling; Diagnostic Test: Mini Mental State Examination (MMSE); Diagnostic Test: Minimal nutritional assessment (MNA-SF); Diagnostic Test: Dual-energy x-ray absorptiometry (DEXA); Device: Dynamometer (Hand grip ); Diagnostic Test: Walking speed
- Control: Elderly patients without sarcopenia
  Interventions: Device: Tongue strength measurement; Procedure: Blood sampling; Diagnostic Test: Mini Mental State Examination (MMSE); Diagnostic Test: Minimal nutritional assessment (MNA-SF); Diagnostic Test: Dual-energy x-ray absorptiometry (DEXA); Device: Dynamometer (Hand grip ); Diagnostic Test: Walking speed

INTERVENTIONS:
Device: Tongue strength measurement — The Iowa Oral Performance Instrument is a validated device for assessing the strength of the tongue. This involves placing the tip of a tube in the mouth and asking the patient to exert pressure on it.
Procedure: Blood sampling — Blood sampling
Diagnostic Test: Mini Mental State Examination (MMSE) — Also called Folstein test, it is an assessment of the patient cognitive and memory functions. It detects cognitive disorders or dementia. The MMSE is quickly realizable and explores several cognitive functions through 30 questions divided into 7 items.
Diagnostic Test: Minimal nutritional assessment (MNA-SF) — The minimal nutritional assessment - short form is a simple, non - invasive and validated scale for the detection of malnutrition in the elderly patient.
Diagnostic Test: Dual-energy x-ray absorptiometry (DEXA) — Dual-energy x-ray absorptiometry (DEXA) is the imaging technique recommended for the diagnosis of sarcopenia.
Device: Dynamometer (Hand grip ) — By placing a dynamometer in the patient's hand and asking him to apply maximum pressure to it, the muscular strength of the extremities of the limbs is estimated.
Diagnostic Test: Walking speed — Walking speed evaluates the muscular performance. The seated patient must get up and walk a distance of 6 meters as quickly as possible without the help of a third party.

SUMMARY:
Sarcopenia is a syndrome characterized by a progressive and generalized loss of skeletal muscle mass, strength and function that increases the risk of physical dependence, impaired quality of life and mortality. This is a major public health problem. Indeed, its prevalence has been estimated at 63.8% for elderly patients hospitalized in acute geriatric unit.

Several methods of sarcopenia screening exist at present. The European Working Group on Sarcopenia in Older People (EWGSOP) proposes to carry out three examinations for the diagnosis of sarcopenia: the Dual-Energy X-ray Absorptiometry (DEXA) test and two motor tests (walking speed and hand test). These measurements have already been evaluated and validated. They are reliable, inexpensive and easily achievable in clinical routine.

Recent studies have shown that decreased muscle mass and / or strength could be associated with dysphagia. Indeed, many muscles of the head and neck are simultaneously solicited for swallowing coordination. This suggests that a reduction in the mass or strength of these muscles could impact the swallowing function. The investigator's hypothesize that loss of lingual muscle strength may be associated with sarcopenia. The study will measure the tongue strength using the Iowa Oral Performance Instrument (IOPI) in a geriatric population with or without sarcopenia.

* Determine the incidence of lingual hypotonia in hospitalized elderly sarcopenia patients.
* To compare the sensitivity, the specificity of the measurement of the force of the tongue with the usual measures proposed by the EWGSOP in the context of screening for sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

Patients hospitalized in an acute geriatric unit within the CHU Brugmann.

Exclusion Criteria:

None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients hospitalized in an acute geriatric unit within the CHU Brugmann.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Tongue strength | 6 months
  The Iowa Oral Performance Instrument is a validated device for assessing the strength of the tongue. This involves placing the tip of a tube in the mouth and asking the patient to exert pressure on it. Thus, a pressure measurement expressed in kPa makes it possible to objectify the tongue strength.

SECONDARY OUTCOMES:
Pre-Albumin concentration | 6 months
  Albumin and pre-albumin are biological markers for undernutrition. Pre-albumin is an earlier marker than albumin because of its shorter half-life, 48 hours versus 21 days. The normal pre-albumin values are between 200 and 400 mg /L, undernutrition is serious if it is less than 150mg/dL.
Albumin concentration | 6 months
  Albumin and pre-albumin are biological markers for undernutrition. Pre-albumin is an earlier marker than albumin because of its shorter half-life, 48 hours versus 21 days.The normal values of albumin are between 40 and 45g/L, between 30 and 35g/L there is moderate undernutrition and under 30g/L it is severe undernutrition.
Mini Mental State Examination (MMSE) score | 6 months
  Also called Folstein test, it is an assessment of the patient cognitive and memory functions. It detects cognitive disorders or dementia. The MMSE is quickly realizable and explores several cognitive functions through 30 questions divided into 7 items: Orientation ability - Learning and transcription skills - Attention and calculation skills - Memory retention capacity - Language and naming capability - Constructive Praxy.
  A MMSE score over 27 indicates normal cognitive functions (maximum: 29). A MMSE score between 24 and 27 indicates mild cognitive impairment. A MMSE score under 24 indicates dementia.
Minimal nutritional assessment (MNA-SF) score | 6 months
  The minimal nutritional assessment - short form is a simple, non - invasive and validated scale for the detection of malnutrition in the elderly patient. It takes into account the patient's loss of appetite, weight loss, motor skills, recent health status, neuropsychological disorders
  The maximum score of the MNA-SF is 14:
  * Greater than or equal to 11: normal nutritional status.
  * Between 8 and 11: risk of malnutrition.
  * Less than 8: proven malnutrition.
Skeletal Mass Muscle Index | 6 months
  Dual-energy x-ray absorptiometry (DEXA) is the imaging technique recommended for the diagnosis of sarcopenia. It gives minimal irradiation and gives an adequate estimate of the appendicular muscle mass (ALM). By dividing the ALM by the size in centimeters, we obtain the Skeletal Mass Muscle Index (SMI). SMI values below 2 standard deviations from the mean point towards sarcopenia.
Hand grip strength | 6 months
  By placing a dynamometer in the patient's hand and asking him to apply maximum pressure to it, the muscular strength of the extremities of the limbs is estimated.
Walking speed | 6 months
  Walking speed evaluates the muscular performance. The seated patient must get up and walk a distance of 6 meters as quickly as possible without the help of a third party. It has been shown that there is a non-linear relationship between walking speed and muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandrine de Buck van Overstraeten, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No